CLINICAL TRIAL: NCT01884337
Title: A Phase IV, Open-Label, Multi-center Study to Evaluate the Safety of Apixaban in Indian Subjects Undergoing Elective Total Knee Replacement or Total Hip Replacement Surgery
Brief Title: Multi-center Study to Evaluate the Safety of Apixaban (BMS-562247) in Indian Subjects Undergoing Elective Total Knee Replacement or Total Hip Replacement Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV185-158
Record Dates: First submitted 2013-06-06; First posted 2013-06-24 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Anticoagulation
MeSH Terms: interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apixaban (2.5 mg) (Experimental): Apixaban 2.5 mg tablets by mouth twice daily, 12 days for TKR subjects or 35 days for THR subjects
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban
  Other Names: Eliquis; BMS-562247

SUMMARY:
The primary purpose of this protocol is to evaluate the safety of Apixaban in prophylaxis of Venous Thromboembolism (VTE) in Indian patients undergoing elective total knee or hip replacement

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Subjects undergoing elective total knee or hip replacement or a revision of at least one component of a total knee or hip replacement

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Known or suspected, acquired or bleeding or coagulation disorder in the subject or a first degree relative
* Active bleeding or at high risk for bleeding.
* Brain, spinal, ophthalmologic, or major surgery or trauma within the past 90 days other than the elective knee/hip surgery
* Active hepatobiliary disease
* Hemoglobin <9 g/dL
* Platelet count <100,000/mm3
* Creatinine clearance <30 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 557 (Actual)
Dates: Start 2015-03-24 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (15):
- India (15):
  - Local Institution, Kozhikode, Kerala
  - Local Institution, Ahmedabad
  - Local Institution, Alappuzha
  - Local Institution, Aurangabad
  - Local Institution, Bangalore
  - Local Institution, Chandigarh
  - Local Institution, Chennai
  - Local Institution, Delhi
  - Local Institution, Hyderabad
  - Local Institution, Kerala
  - Local Institution, Lucknow
  - Local Institution, Mohali
  - Local Institution, Mumbai
  - Local Institution, Nagpur
  - Local Institution, Pune

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in an Indian orthopedic population.
Pre-assignment Details: 557 participants were enrolled, of whom 498 were treated. Of the 59 who were not treated, 42 no longer met study criteria, 6 withdrew consent, 11 due to other reasons. Of the 326 who started Total Knee Replacement, 324 continued into follow-up period and of the 172 who started Total Hip Replacement, 170 continued into follow-up period.
Groups:
- Total Knee Replacement (TKR): Oral administration of apixaban 2.5 mg twice daily (BID) for 2 weeks
- Total Hip Replacement (THR): Oral administration of apixaban 2.5 mg twice daily (BID) for 5 weeks
Period: Treatment
Arm/Group | Total Knee Replacement (TKR) | Total Hip Replacement (THR)
Started | 326 | 172
Continuing Into Follow-up Period | 324 | 171
Completed | 322 | 170
Not Completed | 4 | 2
Not completed — Adverse Event | 2 | 2
Not completed — Subj. request to discont. treatment | 2 | 0
Period: Follow-up Period
Arm/Group | Total Knee Replacement (TKR) | Total Hip Replacement (THR)
Started | 324 | 171
Completed | 323 | 170
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Total Knee Replacement (TKR) | Total Hip Replacement (THR) | Total
Number analyzed (Participants) | 326 | 172 | 498
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (9.59) | 41.7 (13.30) | 54.1 (11.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 237 | 53 | 290
  Male | 89 | 119 | 208
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 9 | 12
  Not Hispanic or Latino | 322 | 163 | 485
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 326 | 172 | 498
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite of International Society on Thrombosis and Haemostasis (ISTH) Major Bleeding/Clinically Relevant Non-major Bleeding (CRNM) While Undergoing Elective TKR or THR at the End of Treatment + 2 Days
Description: TKR = Total knee replacement; THR = Total hip replacement. ISTH major bleeding is 1) Fatal or 2) Bleeding in a critical organ, such as brain, spine, eye, retroperitoneum, joint, heart sac, or skeletal muscle (and resulting in compartment syndrome), or 3) Bleeding that results in a fall of hemoglobin of 2 g/dL or more or transfusion of 2 units or more of packed red cells or whole blood within 24 hours. CRNM bleeding is bleeding that
  1) Is clinically acute and overt 2) Does not satisfy criteria as a major bleed but requires medical intervention, such as a visit to a physician's office, emergency room, or urgent care center for epistaxis
Time Frame: 2 weeks + 2 days for TKR, 5 weeks + 2 days for THR
Population: All participants who received at least one dose of study drug during the Treatment Period
Measure: Count of Participants; unit: Participants
Arm/Group | Total Knee Replacement (TKR) | Total Hip Replacement (THR)
Number analyzed (Participants) | 326 | 172
Participants
  Major Bleeding | 0 | 0
  Clinically Relevant Non-Major Bleeding | 0 | 1
  Major or Clinically Relevant Non-Major Bleeding | 0 | 1
  Any Bleeding | 0 | 1

2. Secondary Outcome: Number of Participants With Composite of Venous Thromboembolism (VTE)/All Cause Death at the End of Treatment + 2 Days
Description: VTE is the combination of deep vein thrombosis and non-fatal pulmonary embolism.
Time Frame: 2 weeks + 2 days for TKR, 5 weeks + 2 days for THR
Population: All participants who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Total Knee Replacement (TKR) | Total Hip Replacement (THR)
Number analyzed (Participants) | 326 | 172
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: AEs are assessed from Day 1 through Day 42 +/- 2 days for Total Knee Replacement Participants; AEs are assessed from Day 1 through Day 65 +/-2 days for Total Hip Replacement Participants.
Arm/Group | TOTAL KNEE REPLACEMENT (TKR) | TOTAL HIP REPLACEMENT (THR)
All-Cause Mortality (participants affected / at risk) | 0/326 | 0/172
Serious Adverse Events (participants affected / at risk) | 2/326 | 0/172
Other Adverse Events (participants affected / at risk) | 23/326 | 6/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TOTAL KNEE REPLACEMENT (TKR) (N=326) | TOTAL HIP REPLACEMENT (THR) (N=172)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TOTAL KNEE REPLACEMENT (TKR) (N=326) | TOTAL HIP REPLACEMENT (THR) (N=172)
Incision site pain (Injury, poisoning and procedural complications) | 23 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2014-07-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT01884337/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT01884337/SAP_001.pdf